CLINICAL TRIAL: NCT07213414
Title: Metagenomic and Metabolomic Analysis Study: Effect of Bifidobacterium Multistrain Probiotic Supplementation on the Abundance and Diversity of Gut Pathogen Microbiota and Levels of Fecal Short Chain Fatty Acid (SCFA) of Preterm Infants in the Neonatal Intensive Care Unit (NICU)
Brief Title: Metagenomic & Metabolomic Study: Bifidobacterium Probiotic Effects on Gut Microbiota & SCFA in Preterm NICU Infants
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Adhariana H. Kaddas, neonatologist, Hasanuddin University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: UH22100576
Record Dates: First submitted 2025-04-14; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Prematurity; Low Birth Weight Neonates
Keywords: Prematurity; Bifidobacterium; Probiotics; Low Birth Weight Neonates
MeSH Terms: conditions — Premature Birth | interventions — Probiotics

STUDY DESIGN:
Masking Description: This study is single-blinded study where the subjects doesn't know if they are included in intervention or comtrol group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-Probiotic Group (No Intervention): The group is for control where the subject would not receive pobiotic intervention.
- Probiotic group (Experimental): The probiotic group is where the subjects received intervention with probiotic suplements one sachet a day.
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — The intervention is giving probiotic supplementation that contains Bifidobacterium longum BB536, Bifidobacterium breve M-16V, Bifidobacterium longum subs.infantis M-63 from Morinaga.
  Arms: Probiotic group

SUMMARY:
One million premature babies die due to prematurity complications, contributing the most to the causes of death in children under 5 years old. Indonesia ranks 5th among countries with the highest premature birth rates in the world, with a mortality rate of 11.1% of all live births, making it the leading cause of neonatal deaths (63.5%). Compared to full-term babies, premature infants are more often born through cesarean section (SC), have an immature immune system, receive antibiotics, and also receive care in the Neonatal Intensive Care Unit (NICU). This can disrupt the formation of gut microbiota early in life. The abnormal bacterial colonization pattern in the intestines of premature infants is dominated by potentially pathogenic microbiota such as Staphylococcus, Klebsiella, Escherichia, and Clostridium. These changes in the gut microbiota ecosystem further increase the risk of severe morbidity during treatment in the NICU, such as necrotizing enterocolitis (NEC), late-onset sepsis (LOS), and long-term morbidities such as asthma and eczema. For decades, probiotics have been researched as non-pathogenic microorganisms that, when given in appropriate amounts, can provide benefits to humans. The results of the research indicate that the administration of probiotics can reduce the incidence of dysbiosis or the imbalance between commensal microbiota and intestinal pathogenic microbiota, strengthen the intestinal barrier, prevent enteropathogenic infections, suppress antimicrobial resistance, increase the body's immunity, and maintain intestinal motility. Based on this mechanism, probiotics are considered to improve outcomes for neonates, especially premature babies. This study was conducted thoroughly through metagenomic and metabolomic analyses of the intestinal microbiota, thereby providing information on the effectiveness of triple strain Bifidobacterium probiotic supplementation based on the abundance of pathogenic and commensal microbiota, alpha and beta diversity, and SCFA levels in the feces of premature infants. The study sample included all accessible populations that met the inclusion criteria. Subjects were randomly divided into two groups: one receiving probiotics and the other not receiving probiotics. Baseline data were collected for all subjects, including their characteristics, anthropometric data, and the antibiotic and probiotic history of mothers and infants. Subsequently, samples were taken from the infants three times, specifically on the first three days (T1), two weeks after probiotic administration (T2), and three weeks after probiotic administration (T3); these samples were then sent to the laboratory for microbiome and metabolomic analysis. The targeted output of this study is the publication of a scientific article in an international journal indexed by Scopus on the analysis of the effect of probiotic administration on metagenomic and metabolomics of the intestinal microbiota of sick premature infants in the NICU. Research on the effectiveness of the triple strain of Bifidobacterium probiotics (Bifidobacterium breve M-16V, Bifidobacterium longum subsp. infantis M-63 and Bifidobacterium longum subsp. longum BB536) in premature infants has never been conducted in South Sulawesi or even in Indonesia. Although research on the effectiveness of the triple strain of Bifidobacterium has been carried out in Japan and Australia, the geographical and ethnic influence on the microbiome pattern is the basis for the need to continue research in Indonesia. So this is certainly a novel value and the results are expected to provide an overview of the microbiome pattern of premature babies in Makassar in particular and in Indonesia in general. In addition, the results of this study can also be the basis for new recommendations regarding the administration of probiotics as an adjunct therapy in the management of premature infants in the NICU.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants (gestational age 28 to <34 weeks) treated in the NICU with a birth weight of 1000 to <2500 grams
* No contraindications to giving the drink in the first 3 days of life
* Parents agree to participate in the study and sign a consent letter.

Exclusion Criteria:

* Major congenital disorders
* Severe sepsis
* No stool production in the first 3 days of life
* Received formula milk that contains probiotics

Ages: 0 Days to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Bifidobacterium Abundance in both groups | This study will include three assessment time points: baseline within the first three days after birth (T1), two weeks after intervention (T2), and immediately before hospital discharge (T3).
  The study compared the abundance of Bifidobacterium genus microbiota between premature infants who received a triple-strain Bifidobacterium probiotic and those who did not.

SECONDARY OUTCOMES:
Klebsiella Abundance in both groups | This study will include three assessment time points: baseline within the first three days after birth (T1), two weeks after intervention (T2), and immediately before hospital discharge (T3).
  The study compared the abundance of potentially pathogenic Klebsiella genus microbiota between premature infants who received a triple-strain Bifidobacterium probiotic and those who did not.
Staphylococcus Abundance in both groups | This study will include three assessment time points: baseline within the first three days after birth (T1), two weeks after intervention (T2), and immediately before hospital discharge (T3).
  The study compared the abundance of potentially pathogenic Staphylococcus genus microbiota between premature infants who received a triple-strain Bifidobacterium probiotic and those who did not.
Alpha Microbiome Diversity | This study will include three assessment time points: baseline within the first three days after birth (T1), two weeks after intervention (T2), and immediately before hospital discharge (T3).
  The study compared alpha microbiome diversity between premature infants who received a triple-strain Bifidobacterium probiotic and those who did not.
Beta Microbiome Diversity | This study will include three assessment time points: baseline within the first three days after birth (T1), two weeks after intervention (T2), and immediately before hospital discharge (T3).
  The study compared microbiome beta diversity between premature infants who received a triple-strain Bifidobacterium probiotic and those who did not.
Total SCFA in both groups | This study will include three assessment time points: baseline within the first three days after birth (T1), two weeks after intervention (T2), and immediately before hospital discharge (T3).
  The study compared the levels of short-chain fatty acids (acetate, butyrate, and propionate) between preterm infants who received a triple-strain Bifidobacterium probiotic and those who did not.
Weight Gain | On birth (baseline) and the day of patient discharged from hospital
  This study will evaluate clinical outcomes to determine the impact of triple-strain Bifidobacterium probiotic supplementation on weight gain.
Hospital Stay Length | From admitted until discharged (during hospitalization)
  This study will evaluate clinical outcomes to determine the impact of triple-strain Bifidobacterium probiotic supplementation on the length of hospital stay.
Duration of Antibiotic Therapy | From admitted until discharged (during hospitalization)
  This study will evaluate clinical outcomes to determine the impact of triple-strain Bifidobacterium probiotic supplementation on the number of days of antibiotic therapy.
Incidence of Necrotizing Enterocolitis | From admitted until discharged (during hospitalization)
  This study will evaluate clinical outcomes to determine the impact of triple-strain Bifidobacterium probiotic supplementation on incidence of necrotizing enterocolitis (NEC)
Incidence of Feeding Intolerance | From admitted until discharged (during hospitalization)
  This study will evaluate clinical outcomes to determine the impact of triple-strain Bifidobacterium probiotic supplementation on the incidence of feeding intolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Adhariana H Kaddas, Neonatologist, Principal Investigator — Child Health Departement, Faculty of Medicine, Hasanuddin University
Locations (3):
- Indonesia (3):
  - Hasanuddin University General Hospital, Makassar, South Sulawesi
  - Dr. Wahidin Sudirohusodo General Hospital, Makassar, South Sulawesi
  - Cahaya Medika General Hospital, Makassar, South Sulawesi

IPD SHARING:
Plan to Share IPD: No
The participant's data will be kept secret to protect the privacy of the participants.

REFERENCES:
- [Background] Takeshita K, Takei H, Tanaka S, Hishiki H, Iijima Y, Ogata H, Fujishiro K, Tominaga T, Konno Y, Iwase Y, Endo M, Ishiwada N, Osone Y, Takemura R, Hamada H, Shimojo N. Effect of multi-strain bifidobacteria supplementation on intestinal microbiota development in low birth weight neonates: a randomized controlled trial. Biosci Microbiota Food Health. 2024;43(4):352-358. doi: 10.12938/bmfh.2023-093. Epub 2024 Jun 17. PMID 39364130